CLINICAL TRIAL: NCT05650203
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of JS009 Monotherapy and JS009 as a Triple Combination Therapy in Combination With Toripalimab and JS006 in Patients With Advanced Malignancies
Brief Title: A Study of JS009 Monotherapy and JS009 as a Triple Combination Therapy in Patients With Advanced Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: the research and develop strategy of Product JS009 adjustment
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS009-002-I
Record Dates: First submitted 2022-11-23; First posted 2022-12-14 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Primary Condition: Advanced Tumors
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS009 as a monotherapy and JS009 Combine with Toripalimab and JS006 (Experimental): 1. JS009 as Monotherapy in first cycle of dose escalation and the triple combination therapy will be administered in subsequent cycles：5 proposed dose levels（18mg, 60mg, 180mg, 600mg, 1200mg).
  2. The triple combination therapy in dose expansion：1 or 2 proposed dose levels, to be determined.
  3. The triple combination therapy in indication expansion：4 or more cohorts, to be determined.
  Interventions: Drug: JS009 as a monotherapy and JS009 as a Triple Combination Therapy in Combination with Toripalimab and JS006

INTERVENTIONS:
Drug: JS009 as a monotherapy and JS009 as a Triple Combination Therapy in Combination with Toripalimab and JS006 — 1. JS009 as Monotherapy in first cycle of dose escalation and as the triple combination therapy will be administered in subsequent cycles：JS009,18mg/60mg/180mg/600mg/1200mg, JS006, fixed dose 600mg, Toripalimab injection fixed dose 240mg,IV infusion, every 3 weeks (q3w).
  2. Triple combination therapy in dose expansion：JS009, 1 or 2 specific dose, with fixed dose of JS006 and Toripalimab Injection, IV infusion, every 3 weeks (q3w).
  3. Triple combination therapy in indication expansion：JS009, 1 specific dose, with fixed dose of JS006 and Toripalimab Injection, IV infusion, every 3 weeks (q3w).

SUMMARY:
The study is being conducted to evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy JS009 as a monotherapy and JS009 as a Triple Combination Therapy in Combination with Toripalimab and JS006 in Patients with Advanced Malignancies, also to explore the RP2D of JS009.

DETAILED DESCRIPTION:
This is an open-label, Phase I study contains dose escalation phase, dose expansion phase and indication expansion phase.

The dose escalation phase will be following the accelerated titration design and the classic 3+3 design, with a planned enrollment of 13 to 30 patients with advanced tumors.

The dose expansion phase will be used safe and tolerable doses, with a planned enrollment of 9 to 24 patients with advanced tumors.

The indication expansion phase will selecte different primary malignancies for investigation of anti-tumor activity. Each Cohort planned to enrollment 20-50 patients with advanced tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign the informed consent form (ICF);
2. Males and females, ≥18 years of age;
3. Histopathology confirmed patients with advanced solid malignancies;
4. Patients who have experienced disease progression on standard therapy, be ineligible for or intolerant of available approved standard therapies known to confer clinical benefit or for whom no effective standard therapy exists; In Indication Expansion Phase, prior tumor types include, but are not limited to:

   * Cohort 1 Non-Small Cell Lung Cancer (NSCLC): patients with locally advanced or metastatic NSCLC, disease recurrence or progression during or after prior therapy with or without anti-PD-(L)1 therapy. The patients must have no known activating EGFR mutations or ALK fusion.
   * Cohort 2 Endometrial Cancer(EC): patients with locally advanced or metastatic EC, disease recurrence or progression during or after prior therapy that included platinum-based chemotherapy.
   * Cohort 3 Ovarian Cancer(OC): patients with locally advanced or metastatic OC, disease recurrence or progression during or after prior therapy that included platinum-based chemotherapy.
   * Cohort 4 Colorectal Cancer(CRC): patients with locally advanced or metastatic CRC, disease recurrence or progression during or after prior therapy with or without anti-PD-(L)1 therapy.
5. In Indication Expansion Phase, prior standard therapy should be ≤ three lines of treatment;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and expected survival ≥12 weeks;
7. At least one measurable lesion per RECISTv1.1; patients without measurable lesions are only acceptable in Dose-Escalation Phase;
8. Agree to provide tumor tissue samples:

   * Freshly prepared sample prior to treatment is recommended, archived sample is acceptable;
   * Applies to dose expansion and indication expansion phases only;
   * Subjects who cannot provide qualified tumor tissue samples may be included with approval from the investigator and the sponsor;
9. Adequate organ and marrow function, as defined below:

   1. Absolute neutrophil count (ANC) ≥ 1.5×109/L (1,500/mm3) with no administration of hematopoietic growth factors for at least 14 days prior to the laboratory evaluations during the screening period; Platelet (PLT) ≥ 100×109/L (100,000/mm3) with no administration of hematopoietic growth factors or platelet transfusions at least 14 days prior to the laboratory evaluations during the screening period;
   2. Hemoglobin (Hb) ≥9 g/dL with no administration of hematopoietic growth factors or red blood cell transfusions for at least 14 days prior to the laboratory evaluations during the screening period;
   3. Total bilirubin (TBIL) < 1.5 × upper limit of normal (ULN);
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN in patients without liver metastases and ALT and AST ≤ 5 × ULN for patients with liver metastases at baseline;
   5. Blood creatinine (Cr) ≤ 1.5 × ULN, or calculated creatinine clearance (Cockcroft-Gault formula) ≥ 50 mL/min, or 24-h urine creatinine clearance ≥ 50 mL/min;
   6. Left ventricular ejection fraction ≥ 50%;
   7. International normalized ratio (INR) ≤ 1.5, and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN except for patients receiving anticoagulation. Patients taking anticoagulants must be on a stable dose and INR or aPTT within the therapeutic goal for warfarin or low molecular weight heparins, respectively for at least 28 days prior to the first dose;
   8. The thyroid function test free triiodothyronine (FT3), free T4 (FT4) and thyroid stimulating hormone (TSH) are within the normal range or no more than Grade 1 abnormalities in patients requiring hormone replacement for those with pre-existing hypothyroidism;
   9. Fridericia-corrected QT interval, ≤ 470 ms for all patients (regardless of sex)
10. Females of childbearing potential who are sexually active with a non-sterilized male partner must agree to use effective contraception Table 1 starting 72 hours before the first dose until 5 months after the final dose, whichever is later. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as at least 12 months with no menses confirmed by FSH levels performed during the screening period);
11. Non-sterilized males who are sexually active with a female partner of childbearing potential must agree to use effective contraception from Day 1 through 5 months after receipt of the final dose.

Exclusion Criteria:

1. Moderate to severe hypersensitivity reaction to toripalimab or other PD-1 blocking antibodies or known allergy to the component of JS009 and JS006 drug product.
2. Prior exposure to antibodies targeting TIGIT, CD112R, CD155, CD113 or related ligands.
3. Concurrent enrollment in another clinical study, or participated in another clinical study within 21 days prior to the first dose of the study drug, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study.
4. Major surgery within 28 days prior to the first dose of the study drug or still recovering from prior surgery.
5. Current or prior use of chemotherapy, radiotherapy, immunotherapy, biologic therapy and targeted therapy within 21 days prior to the first dose of the study drug (Nitrosourea and Mitomycin require 6 weeks interval time between the last dose of chemotherapy and the first dose of the study drug); except： i. The wash-out period for oral medicine is 5 half-lives after discontinuation. ii. The wash-out period is 14 days for palliative radiotherapy (eg. bone radiotherapy to control pain) which has no effect on bone marrow haematopoietic function.

   iii. long-term and stabile hormone therapy. Also, use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
6. Patients with immune-related AEs/SAEs that have led to permanent discontinuation of immune therapies, previously.
7. Current or prior use of immunosuppressive medication within 28 days prior to the first dose of the study drug, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids ≤ 10 mg/day of prednisone or equivalent.
8. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
9. Receipt of live attenuated vaccination within 30 days prior to the first dose of the study drug.
10. Active or prior documented history of another malignancy within 2 years prior to the first dose of the study drug for patients in Dose-Escalation Phase and Dose Expansion Phase, and active or prior documented history of another malignancy within 5 years prior to the first dose of the study drug for patients in Indication Expansion Phase, with the exception of completely cured early-stage malignancies.
11. Symptomatic or untreated central nervous system metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and/or corticosteroids. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 28 days prior to study entry, have no evidence of new or enlarging metastases, and are off steroids.
12. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to baseline or to NCI-CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion and exclusion criteria with the exception of alopecia. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by JS009, toripalimab and/or JS006 may be included (e.g., hearing loss) after consultation with the medical monitor.
13. Active or prior documented autoimmune disease within the past 2 years with the following exceptions: vitiligo, alopecia, endocrinopathies controlled by hormone replacement therapy, rheumatoid arthritis and other arthropathies that have not required immunosuppression other than non-steroidal anti-inflammatory agents, celiac disease controlled by diet, or psoriasis controlled with topical medication.
14. History of primary immunodeficiency.
15. Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, fever of unknown origin that > 38.5°C (patients with neoplastic fever will be evaluated by the investigator for inclusion or exclusion), symptomatic congestive heart failure according to New York Heart Association (NYHA) Functional Classification ≥ Grade 3, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs from JS009, toripalimab and/or JS006, or compromise the ability of the subject to give written informed consent.
16. Known history of active tuberculosis within one year. Has difficulty breathing or current need for continuous oxygen inhalation therapy, or current suffering from active pneumonitis (≥ Grade 2) or interstitial lung disease (except mild radiation pneumonitis).
17. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
18. Patients who are known to be human immunodeficiency virus (HIV) positive.
19. Patients with evidence of hepatitis B or C virus infection, unless their hepatitis is considered to have been cured. (Note that patients with prior hepatitis B virus [HBV] infection must have HBcAb positive, HBsAg negative and have HBV DNA copy number less than the upper limit before study enrollment, and must be treated according to local standards; hepatitis C virus [HCV] infection must have, before study enrollment, negative result of HCV RNA test).
20. Pregnant women. Women who are lactating must agree to discontinue breast-feeding during treatment and for at least 4 months after the last dose of the study drug, whichever is later;
21. Any condition that, in the opinion of the investigator, would interfere with evaluation of JS009, toripalimab and/or JS006 or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | Within the DLT window of the first 2 cycles(42 days) in dose escalation phase
  The Incidence of subjects with adverse event meeting the criteria of dose-limiting toxicity（DLT） in 42 days during dose escalation phase
Incidence and severity of AE as assessed by CTCAE v5.0 | Approximately 2 years.
  The incidence and severity of adverse events (AE)
MTD | Approximately 2 years.
  The highest dose at which no more than 0 of 3 or 1 of 6 patients experienced a DLT during Cycle 1 and 2 during dose escalation phase.
RP2D | Approximately 2 years.
  Recommended phase II dose (RP2D) for JS009 monotherapy and combination therapy

SECONDARY OUTCOMES:
Drug concentration in plasma | Approximately 2 years.
  Drug concentrations including JS009， JS001 and JS006 in individual subjects at different time points after dosing
Immunogenicity | Approximately 2 years.
  Incidence of anti-drug antibody (ADA) and/or neutralizing antibody (Nab), titer of ADA positive samples
ORR | Approximately 2 years.
  Overall Response Rate (ORR) was assessed based on RECIST V1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yilong WU, Ph.D, Study Chair — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No